CLINICAL TRIAL: NCT00964665
Title: A Pharmacokinetic/Pharmacodynamic Evaluation of ABF656 in Subjects With Chronic Hepatitis B, e Ag+, Infection.
Brief Title: Pharmacokinetic/Pharmacodynamic of Albinterferon Alfa-2b in Chronic Hepatitis B, eAg+, Infection Subjects
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABF656A2206; EudraCT 2008-006933-29
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B,; Chronic,; Hepatitis B e Antigens positive
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Bronchiolitis Obliterans Syndrome | interventions — albinterferon alfa-2b; peginterferon alfa-2a

ARMS (5):
- Group 1 ABF656 900ug Q2w (Experimental)
  Interventions: Drug: albinterferon alfa-2b
- Group 2 ABF656 900ug Q4w (Experimental)
  Interventions: Drug: albinterferon alfa-2b
- Group 3 AB656 1200ug Q4w (Experimental)
  Interventions: Drug: albinterferon alfa-2b
- Group 4 ABF656 1500ug Q4w (Experimental)
  Interventions: Drug: albinterferon alfa-2b
- Group 5 Pegasys® 180µg qw (Active Comparator)
  Interventions: Drug: Pegasys®

INTERVENTIONS:
Drug: albinterferon alfa-2b
  Arms: Group 1 ABF656 900ug Q2w
Drug: albinterferon alfa-2b
  Arms: Group 2 ABF656 900ug Q4w
Drug: albinterferon alfa-2b
  Arms: Group 3 AB656 1200ug Q4w
Drug: albinterferon alfa-2b
  Arms: Group 4 ABF656 1500ug Q4w
Drug: Pegasys®
  Arms: Group 5 Pegasys® 180µg qw

SUMMARY:
This study will assess the efficacy of ABF656 in chronic hepatitis B characterized by HBeAg positivity. The study is designed to establish a dose response and safety relationship sufficient to allow the subsequent design and conduct of Phase 3 trials. The trial is also designed to generate the PK data in hepatitis B patients to satisfy regulatory requirements in China.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years of either non-child bearing potential or if of child bearing potential on two adequate forms of birth control
* Chronic HBV infection (serum HBsAg detectable for > 6 months)
* Serum HBeAg positive with HBV DNA >106copies/mL (or >200,000 IU/mL)
* Serum ALT must be > 2 x ULN but below 10 x ULN

Exclusion Criteria:

* Steroid treatment or immunosuppression 3 months prior to entry.
* Chest X-ray with clinically significant active inflammatory process, history of significant pulmonary disease or any history of interstitial lung disease.
* Hb< 10g/dL or, and ANC < 750/mm3 or , and platelet count < 75,000 mm3 .
* Significant chronic medical conditions other than chronic hepatitis B which in the opinion of the investigator preclude enrollment into the study.
* Evidence of hepatic decompensation (i.e., Child-Pugh score of B or C).
* Seropositive for HIV, HCV, or HDV (Hepatitis Delta virus).
* History of hypothyroidism or current treatment for thyroid disease.
* Patients with treated or untreated malignancy of any organs, with the exception of localized basal cell carcinoma

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety, tolerability and pharmacodynamic effect of various doses of albinterferon alfa-2b in hepatitis B patients on seroconversion of hepatitis markers. Measure: Clinical laboratory. HBV DNA level and HBeAg seroconversion rate. | 48 weeks

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics at different doses of albinterferon alfa-2b in patients with chronic hepatitis B infection. Measure: Serum concentration of albinterferon alfa-2b | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Institute for BioMedical Research
Locations (12):
- Novartis Investigator Site, Beijing, China
- Hong Kong (2):
  - Novartis Investigator Site, Shatin
  - Novartis Investigator Site, Taipo
- Poland (3):
  - Novartis Investigator Site, Bialystok
  - Novartis Investigator Site, Lodz
  - Novartis Investigator Site, Warsaw
- Taiwan (3):
  - Novartis Investigator Site, Kaohsiung City
  - Novartis Investigator Site, Taipei
  - Novartis Investigator Site, Tau-Yuan County
- Thailand (3):
  - Novartis Investigator Site, Bangkok
  - Novartis Investigator Site, Chiang Mai
  - Novartis Investigator Site, Songkhla

REFERENCES:
- [Background] Cooksley WG, Piratvisuth T, Lee SD, Mahachai V, Chao YC, Tanwandee T, Chutaputti A, Chang WY, Zahm FE, Pluck N. Peginterferon alpha-2a (40 kDa): an advance in the treatment of hepatitis B e antigen-positive chronic hepatitis B. J Viral Hepat. 2003 Jul;10(4):298-305. doi: 10.1046/j.1365-2893.2003.00450.x. PMID 12823597
- [Derived] Colvin RA, Tanwandee T, Piratvisuth T, Thongsawat S, Hui AJ, Zhang H, Ren H, Chen PJ, Chuang WL, Sobhonslidsuk A, Li R, Qi Y, Praestgaard J, Han Y, Xu J, Stein DS; ABF656A2206 Study Group. Randomized, controlled pharmacokinetic and pharmacodynamic evaluation of albinterferon in patients with chronic hepatitis B infection. J Gastroenterol Hepatol. 2015 Jan;30(1):184-91. doi: 10.1111/jgh.12671. PMID 24995515